CLINICAL TRIAL: NCT04559711
Title: Demonstration Programme to Improve Maternal Nutrition Service Delivery Including Multiple Micronutrient Supplementation (MMS) Through Public Health ANC Platforms: A Community Based Cluster Randomized Control Trial
Brief Title: cRCT to Improve Maternal Nutrition Service Delivery During ANC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: UNICEF (Other); Penn State University (Other); Government of Bangladesh (Other Government); World Bank (Other); Sight and Life, Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-19124
Record Dates: First submitted 2020-09-06; First posted 2020-09-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Maternal Nutritional Deficiency During Childbirth
Keywords: Maternal nutrition; Antenatal care; Randomized control trial; Multiple micro-nutrient supplementation; Bangladesh

STUDY DESIGN:
Intervention Model Description: Two parallel arm superiority community based cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Strengthening coverage and quality of nutrition services including MMS during ANC
  Interventions: Other: Strengthening coverage and quality of nutrition services during ANC
- Comparison arm (No Intervention): Existing provision of nutrition services during ANC.

INTERVENTIONS:
Other: Strengthening coverage and quality of nutrition services during ANC — Intervention clusters will receive inputs both at facility level and community level. The supply side inputs will include efforts for improving facility readiness, quality of nutrition services during ANC, multiple micronutrient supplementation(MMS) and strengthening monitoring and supervision for ANC. On the other hand, community mobilization interventions will be carried out for demand creation. All public health facilities providing ANC services in the intervention area will be included; Union Health & Family Welfare Center, Community Clinic and Satellite Clinic.
  Arms: Intervention arm

SUMMARY:
Malnutrition among women of reproductive age is a significant public health problem in Bangladesh, with major implications for a woman's own health and that of her newborn child. The principal drivers for maternal malnutrition in Bangladesh are poor-quality diets, care seeking practices and access to health care. An ideal contact point for pregnant women are antenatal care visits (ANC). However, the provision of maternal nutrition services through government systems is inadequate with just 29% of pregnant women attending all 4 ANC visits and 18% of women consuming at least 100 IFA tablets. Moreover, WHO made a context specific recommendation that countries with a high prevalence of nutritional deficiencies may choose to adopt multiple micronutrient supplementation (MMS) over iron folic acid (IFA). The health benefits of MMS cannot be harnessed without a properly functioning delivery platform. A multifaceted approach focusing on improving the quality of ANC, the supply system for these services, engagement with communities, in addition to the adoption of MMS may have large benefits to women and children in Bangladesh. UNICEF and the Bill and Melinda Gates Foundation have partnered with several different organizations, including the GoB, Sight & Life, Pennsylvania State University (PSU) and icddr, b to design and assess outcome of a community based randomized control trial to improve coverage and quality of maternal nutrition service delivery through ANC platform. The investigators hypothesize that implementation of demonstration programme will result in 60% relative improvement in the coverage of 100+ MMS among women who received 4+ANC in the intervention areas compared to the coverage of 100+ IFA among women who received 4+ANC in comparison areas.

DETAILED DESCRIPTION:
1. Burden:

   Globally, it is recognized that pre-conception and during pregnancy malnutrition among women is an underlying cause of maternal morbidity, mortality, and poor birth outcomes including low birth weight babies. In Bangladesh, the poor pre-conception and pregnancy nutritional status of women contributes to the prevailing high rates of low birth weight among newborns. Each year, approximately 860,000 or 28% of babies are born with low birth weight (<2500g) greatly increasing their risk of stunting and wasting, and diet-related non-communicable diseases in adult life.
2. Knowledge gap:

   An ideal contact point for pregnant women for delivering nutrition services are antenatal care visits (ANC). However, the provision of maternal nutrition services through government systems is inadequate in terms of coverage and quality. Overall 29% of pregnant women in Bangladesh receive 4 ANC and 18% of women consume at least 100 IFA tablets. Moreover recent WHO context specific recommendation suggest countries with a high prevalence of nutritional deficiencies may choose to adopt multiple micronutrient supplementation (MMS) over iron folic acid (IFA). The health benefits of MMS cannot be harnessed without a properly functioning delivery platform. A multifaceted approach focusing on improving the quality of ANC, the supply system for these services, engagement with communities, in addition to the adoption of MMS may have large benefits to women and children in Bangladesh. UNICEF and the Bill and Melinda Gates Foundation have partnered with several different organizations, including the GoB and icddr, b to build a comprehensive understanding of where gaps in ANC and nutritional care delivery currently exist, how to bridge these gaps, strengthen both the supply and service system, engage with a larger number of pregnant women, and finally encourage the adoption of the programme across Bangladesh.
3. Relevance:

The most recent State of Food Security and Nutrition in Bangladesh Report found that 66% of women did not consume adequately diversified diets, indicating micronutrient deficiencies. A growing body of evidence has found that multiple micronutrient supplementation (MMS) may result in better neonatal outcomes for undernourished pregnant women. MMS has been associated with reductions in the number of LBW and small for gestational age (SGA) births, as well as a reduction in the number of preterm births among mothers who were underweight in both meta-analysis and a randomized control trial in Bangladesh. Recently in Dhaka, Bangladesh national anaemia consultation workshop was held, which also recommended changing the formulation from IFA only to a multi-micronutrient supplement for pregnant women and to scale up providing children with MNPs.

Objectives:

The study will be conducted in two phases. The specific objectives are;

Phase I:

1. To conduct a comprehensive situation analysis to identify gaps in the existing maternal nutrition service delivery and coverage of maternal nutrition interventions
2. To conduct a formative research to inform design of a demonstration programme improving maternal nutrition service delivery through public health ANC platforms

   Phase II:
3. To implement a two parallel arm superiority community based cluster randomized controlled trial (cRCT) to assess whether implementation of the demonstration programme improves coverage and quality of nutrition service delivery through public health ANC platforms

Methods:

During phase I,a comprehensive situation analysis and a formative research will be conducted to inform the design of a demonstration programme improving maternal nutrition service delivery through public health ANC platforms. The study will employ a quantitative approach for comprehensive situation analysis involving health facility assessment, health care provider interviews, ANC observation, exit interviews of the women receiving ANC and household hold survey. The situation analysis will enable the investigators to identify the gaps of in terms of coverage and quality of maternal nutrition services through public health ANC platforms, knowledge, attitude and practices of the health care providers and pregnant women regarding maternal nutrition. A formative research will be conducted to inform the design of the demonstration programme. Demonstration programme will be designed based on the findings from the baseline situation analysis and formative research. During Phase II, a two parallel arm superiority community based cluster randomized control trial (cRCT) will be implemented to assess whether implementation of the demonstration programme improves coverage and quality of Nutrition services through public health ANC platforms. Unit of randomization will be unions. A total of 40 unions will be selected from two districts and paired based on principle component analysis (PCA) score. PCA will take into consideration coverage of ANC and IFA and socio-demographics characteristics (literacy rate, provision of pure drinking water, sanitation facilities). Later each of the pair will be randomized into either intervention or comparison arm. Cross sectional surveys will be conducted to assess coverage of key maternal health and nutrition indicators. Additionally a cohort of pregnant women from intervention and comparison facilities will be followed to measure the change in quality of nutrition service delivery and consumption of 100+ MMS tablets during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women coming for ANC in the public health facilities
* Provide consent to participate in the study

Exclusion Criteria:

* pregnant women who will not provide consent to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 2520 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the coverage of 100+ MMS supplementation among recently delivered women who received 4 ANC from the baseline to the end of the project in the intervention and the comparison areas | Baseline (0 months) and end of project (18 months)
  Change in the proportion of pregnant women received at least 4 ANCs and consumed 100+ MMS supplementation in their last pregnancy from baseline to the end of the project in intervention and comparison areas

SECONDARY OUTCOMES:
Change in the quality of nutrition services during ANC (4 ANC MMS/IFA, weight gain monitoring and dietary counseling) from the baseline to the end of the project in the intervention and the comparison areas | Baseline (0 months) and end of project(18 months)
  Change in the proportion of recently delivered women attended at least 4 ANCs and received three maternal nutrition services (MMS/IFA, weight gain monitoring and dietary counseling) from the baseline to the end of the project in the intervention and the comparison areas
Change in the coverage of 4+ ANC from the baseline to the end of the project in the intervention and the comparison areas | Baseline (0 months) and end of project(18 months)
  Change in the proportion of recently delivered women who received at least 4 ANC in their last pregnancy from the baseline to the end of the project in the intervention and the comparison areas
Change in the coverage of nutrition counselling from the baseline to the end of the project in the intervention and the comparison areas | Baseline (0 months) and end of project(18 months)
  Change in the proportion of recently delivered women who received nutrition counselling (diet, supplement & lifestyle) in their last pregnancy from the baseline to the end of the project in the intervention and the comparison areas
Change in the coverage of weight monitoring from the baseline to the end of the project in the intervention and the comparison areas | Baseline (0 months) and end of project(18 months)
  Change in the proportion of recently delivered women who received at least 4 ANC and whose weight was recorded in the ANC card/ register for all four ANCs in their last pregnancy from the baseline to the end of the project in the intervention and the comparison areas

CONTACTS AND LOCATIONS:
Overall Officials: Sk Masum Billah, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Bogra, Bangladesh